CLINICAL TRIAL: NCT05634915
Title: Clinical Study of rATG Individualized Administration for Prevention of GVHD and Maintenance of GVL in Haploidentical Hematopoietic Stem Cell Transplantation.
Brief Title: Clinical Study of rATG Individualized Administration in Haploidentical Hematopoietic Stem Cell Transplantation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ATGIA2022
Record Dates: First submitted 2022-11-22; First posted 2022-12-02 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2022-11

CONDITIONS: Hematopoietic Stem Cell Transplantation; Acute Leukemia
Keywords: Antithymocyte Globulin; Population pharmacokinetic model; Haploidentical Hematopoietic Stem Cell Transplantation; Acute Leukemia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Individual dose of ATG (Experimental): The total individual ATG dose was calculated based on population pharmacokinetic modeling. ATG was intravenously infused every day from day -5 to day -2.
  Interventions: Drug: Individual ATG
- ATG 10mg/kg (Active Comparator): The total ATG dose was 10mg/kg. ATG was intravenously infused every day from day -5 to day -2.
  Interventions: Drug: ATG

INTERVENTIONS:
Drug: Individual ATG — Individual dose of ATG: Individual dose of ATG was Intravenous infused every day from day -5 to day -2 (total ATG dose was calculated based on population pharmacokinetic modeling). Prophylaxis against graft-versus-host disease (GVHD) was performed with cyclosporine A, mycophenolate mofetil, and low-dose methotrexate.
  Arms: Individual dose of ATG
Drug: ATG — ATG 10mg/kg: The total ATG dose was 10mg/kg. ATG was intravenously infused every day from day -5 to day -2. Prophylaxis against graft-versus-host disease (GVHD) was performed with cyclosporine A, mycophenolate mofetil, and low-dose methotrexate.
  Arms: ATG 10mg/kg

SUMMARY:
The purpose of this prospective, open-label, pairing design, single-center study is to evaluate the effect of individualized rATG dosing vs traditional weight-based rATG dosing regimen（10mg/kg）for patients with acute leukemia undergoing a myeloablative conditioning regimen and haploidentical hematopoietic stem cell transplantation (haplo-HSCT).

DETAILED DESCRIPTION:
Allogeneic hematopoietic stem-cell transplantation (HSCT) is a potentially curative treatment option for acute leukemia. Haploidentical hematopoietic stem cell transplantation (haplo-HSCT) has become the main choice for acute leukemia in China. Major difficulties of the procedure include graft-versus-host disease (GVHD), graft failure, and relapse. As an important role of haplo-HSCT, Rabbit anti-thymocyte globulin (rATG), a polyclonal rabbit-derived antibody that depletes lymphocytes, including T cells, was introduced to prevent GVHD and transplant rejection.

The recommended dose of rATG in haplo-HSCT is 10 mg/kg. However, while the traditional weight-based rATG dosing regimen (10mg/kg) reduces the incidence of GVHD, it increases the risk of delayed immune reconstitution, viral reactivation, and relapse in patients. Our previous retrospective study showed that active ATG exposure (area under the curve, AUC)) post-transplantation is associated with immune reconstitution, GVHD, relapse, survival, and viral reactivation in HSCT of acute leukemia patients. Identifying the optimal dose of ATG to achieve the optimal exposure range of active ATG is a pressing clinical issue.

The pharmacokinetics of ATG varies significantly in both pediatric and adult populations, especially the active ATG levels, and clarifying the relationship between the pharmacokinetics of ATG and the prognosis of patient outcomes can help in precise treatment. By constructing a population pharmacokinetic model of ATG, we can provide an individualized optimal dose of ATG based on factors prior to transplantation. ATG individualized administration may improve the survival and quality of life of patients undergoing haplo-HSCT. A prospective pairing design trial is required to evaluate the effect of individualized rATG dosing vs traditional weight-based rATG dosing regimen (10mg/kg) for patients with acute leukemia undergoing haplo-HSCT.

ELIGIBILITY:
Inclusion Criteria:

1. All patients were diagnosed with acute leukemia.
2. All patients should have the indication of Haploidentical hematopoietic stem cell transplant and receive the myeloablative conditioning regimen.
3. All patients should sign an informed consent document indicating that they understand the purpose of and procedures required for the study and be willing to participate in the study.

Exclusion Criteria:

Patients with any conditions not suitable for the trial (investigators' decision).

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-12-20 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Cumulative incidences of aGVHD | 100 days after transplantation
  The diagnosis and grading of aGVHD are based on the modified Glucksberg grading standard.
CD4+ immune reconstitution | 3 months after transplantation
  CD4+ T-cells >0·05 × 10⁹/L twice within 3 months after transplantation
Leukemia-free survival (LFS) | 1 years after transplantation
  Leukemia-free survival (LFS) is defined as the time from enrollment to relapse of primary disease or death from any cause, whichever occurred first.

SECONDARY OUTCOMES:
Cumulative incidences of cGVHD | 1 years after transplantation
  Chronic GVHD can be classified as "limited" or "extensive" according to the Seattle criteria, and also be classified as "mild" or "moderate" or "severe" according to the National Institutes of Health (NIH) criteria.
Cumulative incidences of EBV reactivation | 1 years after transplantation
  The cumulative incidences of EBV reactivation after transplantation
Cumulative incidence of CMV reactivation | 1 years after transplantation
  The cumulative incidences of CMV reactivation after transplantation.
Neutrophil engraftment | 1 month after transplantation
  Neutrophil engraftment is defined as the first of 3 consecutive days with an absolute neutrophil count > 0.5 × 10^9/L.
Platelet engraftment | 1 month after transplantation
  Platelet engraftment is defined as the first of 7 consecutive days with an absolute platelet count > 20 × 10^9/L independent from transfusion.
Overall survival (OS) | 1 years after transplantation
  Overall survival (OS) is defined as the time from randomization to death resulting from any cause.
GVHD-free and relapse-free survival (GRFS) | 1 years after transplantation
  GRFS is defined as the time from graft infusion to the onset of grades 3 to 4 aGVHD, moderate to severe cGVHD, or relapse/disease progression/death.
Non-relapse mortality (NRM) | 1 years after transplantation
  Non-relapse mortality (NRM) is defined as the time from enrollment to death of any causes other than hematologic disease relapse.
Relapse-related mortality (RRM) | 1 years after transplantation
  Relapse-related mortality (RRM) is defined as the time from enrollment to death of relapse.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaowen Tang, PhD, Study Chair — The First Affiliated Hospital of Soochow University
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China